CLINICAL TRIAL: NCT03381872
Title: Randomized Controlled Trial of Intravascular Imaging Guidance Versus Angiography-Guidance on Clinical Outcomes After Complex Percutaneous Coronary Intervention (RENOVATE-COMPLEX-PCI)
Brief Title: Intravascular Imaging- Versus Angiography-Guided Percutaneous Coronary Intervention For Complex Coronary Artery Disease
Acronym: RENOVATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Renovate16453143
Record Dates: First submitted 2017-12-16; First posted 2017-12-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Intravascular Imaging; Intravascular Ultrasound; Optical Coherence Tomography; Complex Lesion; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Percutaneous Coronary Intervention; Drug-Eluting Stents; Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Prospective, open label, two-arm, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: All end points will be independently adjudicated by Clinical Event Adjudication Committee (CEAC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular imaging arm (Active Comparator): The choice of intravascular imaging devices such as IVUS or OCT during PCI will be left to the operator's discretion. In case of staged procedure during the same hospitalization, following the initially allocated strategy would be strongly recommended. Use of intravascular imaging devices will be allowed at any step of PCI (pre-PCI, during PCI and post-PCI), but intravascular imaging evaluation after stent implantation will be mandatory.
  Interventions: Procedure: Percutaneous coronary intervention for complex lesion; Device: Drug-eluting stent; Device: Intravascular imaging (IVUS or OCT); Device: Drug-coated balloon
- Angiography arm (Active Comparator): The PCI procedure in this group will be performed as standard procedure. After deployment of stent, stent optimization will be done based on angiographic findings. The optimization guided by angiography should meet the criteria of angiographic residual diameter stenosis less than 10% by visual estimation and the absence of flow limiting dissection (≥Type C dissection). When angiographic under-expansion of the stent is suspected, adjunctive balloon dilatation will be strongly recommended. In case of staged procedure during the same hospitalization, following the initially allocated strategy would be strongly recommended.
  Interventions: Procedure: Percutaneous coronary intervention for complex lesion; Device: Drug-eluting stent; Device: Drug-coated balloon

INTERVENTIONS:
Procedure: Percutaneous coronary intervention for complex lesion — In patients who have complex coronary lesions, PCI will performed using intravascular imaging or angiography only according to the allocated arms
  1. Intravascular imaging arm
  2. Angiography arm
     * Definition of Complex Lesions
       1. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) with side branch ≥2.5mm size
       2. Chronic total occlusion (≥3 months) as target lesion
       3. PCI for unprotected left main (LM) disease (LM os, body, distal LM bifurcation including non-true bifurcation)
       4. Implanted stent length ≥38mm
       5. Multi-vessel PCI (≥2 major epicardial coronary arteries treated at one PCI session)
       6. Multiple stent needed (≥3 more stent per patient)
       7. In-stent restenosis lesion as target lesion
       8. Severely calcified lesion (encircling calcium in angiography)
       9. Ostial coronary lesion (LAD, LCX, RCA)
Device: Drug-eluting stent — All patient will be received percutaneous coronary intervention with second generation drug-eluting stent or drug-coated balloon.
Device: Intravascular imaging (IVUS or OCT) — IVUS Reference site: Largest lumen, Plaque burden <50% Stent sizing: By measuring vessel diameter (external elastic membrane) at proximal and distal reference sites. The averaged value of the proximal and distal reference external elastic membrane diameter will be used as stent diameter
  OCT Reference site: Most normal looking segment, No Lipidic plaque Stent sizing: [1] By measuring vessel diameter at the distal reference sites (in case of ≥180° of the external elastic membrane can be identified). In this case, stent diameter will be determined using mean external elastic membrane diameter at the distal reference, rounded down to the nearest 0.25 mm.
  [2] By measuring lumen diameter at the distal reference sites (in case of ≥180° of the external elastic membrane cannot be identified). In this case, stent diameter will be determined using mean lumen diameter at the distal reference, rounded up to the nearest 0.25 mm.
  Arms: Intravascular imaging arm
Device: Drug-coated balloon — All patient will be received percutaneous coronary intervention with second generation drug-eluting stent or drug-coated balloon.

SUMMARY:
The aim of the study is to compare clinical outcomes between intravascular imaging-guided versus angiography-guided percutaneous coronary intervention (PCI) in complex lesions.

DETAILED DESCRIPTION:
After introduction of the 2nd generation drug-eluting stents (DES), the rates of device-related failure or target lesion failure such as restenosis and stent thrombosis has been markedly decreased, compared with the era of bare metal stents or 1st generation DES. Nevertheless, patients undergoing percutaneous coronary intervention (PCI) for complex lesions, for example, chronic total occlusion (CTO), left main disease, true bifurcation lesion, long lesion, multi-vessel PCI, multiple overlapping stents, or severely calcified lesions have significantly worse clinical outcomes than those with non-complex lesions.

During the PCI procedure, intravascular ultrasound (IVUS) and optical coherence tomography (OCT) are useful tools for providing information on preintervention lesion characteristics, including vulnerable plaques, lesion severity, length, and morphology; on postintervention optimal stent implantation for stent expansion, extension, and apposition; and on possible complications after stent implantation. Therefore, intravascular imaging guidance may improve clinical outcomes after complex PCI. However, although previous randomized controlled trial (RCT) and registries showed significantly lower rates of major adverse clinical events following IVUS-guided PCI compared with angiography-guided PCI, the RCTs were limited with small sample size and dealt with very selected lesion subsets such as CTO or long lesion. Moreover, it is uncertain whether OCT-guided PCI improves clinical outcomes compared with angiography-guided PCI. Meanwhile, appropriate imaging modality may differ according to patient and lesion characteristics.

One of the ways to maximize the advantage of intravascular imaging is choice of intravascular imaging devices by the operator's discretion. Therefore, the current RENOVATE-COMPLEX-PCI (Randomized Controlled Trial of Intravascular Imaging Guidance versus Angiography-Guidance on Clinical Outcomes After Complex Percutaneous Coronary Intervention) is designed to investigate whether PCI under guidance of intravascular imaging devices (IVUS or OCT) chosen by operators would improve clinical outcomes compared with angiography-guided PCI in patients with complex lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥19 years old
* Coronary artery disease requiring PCI
* Patients with complex lesion

  1. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) with side branch ≥2.5mm size
  2. Chronic total occlusion (≥3 months) as target lesion
  3. Unprotected LM disease PCI (LM ostium, body, distal LM bifurcation including non-true bifurcation)
  4. Long coronary lesions (implanted stent ≥38 mm in length)
  5. Multi-vessel PCI (≥2 vessels treated at one PCI session)
  6. Multiple stents needed (≥3 more stent per patient)
  7. In-stent restenosis lesion as target lesion
  8. Severely calcified lesion (encircling calcium in angiography)
  9. Ostial coronary lesion (LAD, LCX, RCA)
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Target lesions not amenable for PCI by operators' decision
* Cardiogenic shock (Killip class IV) at presentation
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, or Everolimus
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Pregnancy or breast feeding
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1639 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vessel Failure | 1-year after last patient enrollment
  A composite of cardiac death, target vessel MI, and clinically-driven target vessel revascularization

SECONDARY OUTCOMES:
Target vessel failure without procedure-related MI | 1-year after last patient enrollment
  A composite of cardiac death, spontaneous target vessel MI, and clinically-driven target vessel revascularization
Cardiac death or target-vessel related MI | 1-year after last patient enrollment
  Cardiac death or target-vessel related MI
All-cause death | 1-year after last patient enrollment
  any death
Cardiac death | 1-year after last patient enrollment
  cardiac death
Target vessel MI with procedure-related MI | 1-year after last patient enrollment
  Target vessel MI with procedure-related MI
Target vessel MI without procedure-related MI | 1-year after last patient enrollment
  Target vessel MI without procedure-related MI
Any MI with procedure-related MI | 1-year after last patient enrollment
  Any MI with procedure-related MI
Any MI without procedure-related MI | 1-year after last patient enrollment
  Any MI without procedure-related MI
Non-target vessel related MI | 1-year after last patient enrollment
  Non-target vessel related MI
Target lesion revascularization | 1-year after last patient enrollment
  TLR
Target vessel revascularization | 1-year after last patient enrollment
  TVR
Any revascularization | 1-year after last patient enrollment
  clinically-driven revascularization
Stent thrombosis | 1-year after last patient enrollment
  definite stent thrombosis
Incidence of contrast-induced nephropathy | 48-72 hours after index procedure
  CIN was defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline within 48-72 hours after contrast agent exposure
Total amount of contrast use | Immediate after index procedure
  Total amount of contrast use during index hospitalization
Total procedure time | Immediate after index procedure
  Total procedure time during index hospitalization
Total medical cost | 1-year after last patient enrollment
  Total medical cost
Target vessel Failure | 4 years after last patient enrollment
  A composite of cardiac death, target vessel MI, and clinically-driven target vessel revascularization
Target vessel failure without procedure-related MI | 4 years after last patient enrollment
  A composite of cardiac death, spontaneous target vessel MI, and clinically-driven target vessel revascularization
All-cause death | 4 years after last patient enrollment
  any death
Cardiac death | 4 years after last patient enrollment
  cardiac death
Target vessel MI with procedure-related MI | 4 years after last patient enrollment
  Target vessel MI with procedure-related MI
Target vessel MI without procedure-related MI | 4 years after last patient enrollment
  Target vessel MI without procedure-related MI
Any MI with procedure-related MI | 4 years after last patient enrollment
  Any MI with procedure-related MI
Any MI without procedure-related MI | 4 years after last patient enrollment
  Any MI without procedure-related MI
Non-target vessel related MI | 4 years after last patient enrollment
  Non-target vessel related MI
Target lesion revascularization | 4 years after last patient enrollment
  TLR
Target vessel revascularization | 4 years after last patient enrollment
  TVR
Any revascularization | 4 years after last patient enrollment
  clinically-driven revascularization
Stent thrombosis | 4 years after last patient enrollment
  definite stent thrombosis
Bleeding (BARC definition) | 4 years after last patient enrollment
  BARC Classification (2,3, or 5)
Bleeding (TIMI definition) | 4 years after last patient enrollment
  TIMI Classification (Minimal, Minor, Major)

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked

REFERENCES:
- [Derived] Jo J, Lee SY, Kwon W, Lee SJ, Lee JY, Lee SH, Shin D, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Choi KH, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Lee SY, Lee JM; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided Versus Angiography-Guided Complex PCI in Patients With High Bleeding Risk: A Secondary Analysis of the RENOVATE-COMPLEX PCI Trial. Circ Cardiovasc Interv. 2025 Mar;18(3):e014952. doi: 10.1161/CIRCINTERVENTIONS.124.014952. Epub 2025 Mar 18. PMID 40100948
- [Derived] Lee JM, Lee SY, Kwon W, Lee SJ, Lee JY, Lee SH, Shin D, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Choi KH, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging Predictors Associated With Cardiovascular Events After Complex PCIs. Circ Cardiovasc Interv. 2025 Feb;18(2):e014920. doi: 10.1161/CIRCINTERVENTIONS.124.014920. Epub 2025 Feb 18. PMID 39965046
- [Derived] Lee SY, Lee SJ, Kwon W, Lee SH, Shin D, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Choi KH, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Lee JY, Lee JM, Investigators TR. Outcomes of intravascular imaging-guided percutaneous coronary intervention according to lesion complexity. EuroIntervention. 2025 Feb 3;21(3):e171-e182. doi: 10.4244/EIJ-D-24-00755. PMID 39901632
- [Derived] Hong D, Ha J, Choi KH, Lee SH, Shin D, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Park TK, Lee JM; RENOVATE-COMPLEX-PCI Investigators. Prognostic impact of intravascular imaging in percutaneous coronary intervention according to atherothrombotic risk: a post hoc analysis of a randomized clinical trial. Rev Esp Cardiol (Engl Ed). 2025 Jun;78(6):542-552. doi: 10.1016/j.rec.2024.11.007. Epub 2024 Dec 4. English, Spanish. PMID 39643207
- [Derived] Choi KH, Park TK, Song YB, Lee JM, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Yoon HJ, Park YH, Lee WS, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Yang JH, Choi SH, Gwon HC, Hahn JY, Nam CW; RENOVATE COMPLEX-PCI Investigators. Intravascular Imaging and Angiography Guidance in Complex Percutaneous Coronary Intervention Among Patients With Diabetes: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417613. doi: 10.1001/jamanetworkopen.2024.17613. PMID 38913377
- [Derived] Lee SY, Choi KH, Kim CJ, Lee JM, Song YB, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Jeong JO, Song PS, Kim SE, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY; RENOVATE-COMPLEX-PCI Investigators. Impact of Intravascular Imaging-Guided Stent Optimization According to Clinical Presentation in Patients Undergoing Complex PCI. JACC Cardiovasc Interv. 2024 May 27;17(10):1231-1243. doi: 10.1016/j.jcin.2024.03.021. PMID 38811104
- [Derived] Cha JH, Lee JM, Choi KH, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY, Lee WS, Song YB; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided Optimization of Complex Percutaneous Coronary Intervention by Sex: A Subgroup Analysis of the RENOVATE-COMPLEX-PCI Trial. JAMA Cardiol. 2024 May 1;9(5):466-474. doi: 10.1001/jamacardio.2024.0291. PMID 38568686
- [Derived] Hong D, Lee J, Lee H, Cho J, Guallar E, Choi KH, Lee SH, Shin D, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Kang D, Lee JM; RENOVATE-COMPLEX-PCI Investigators. Cost-Effectiveness of Intravascular Imaging-Guided Complex PCI: Prespecified Analysis of RENOVATE-COMPLEX-PCI Trial. Circ Cardiovasc Qual Outcomes. 2024 Mar;17(3):e010230. doi: 10.1161/CIRCOUTCOMES.123.010230. Epub 2024 Mar 13. PMID 38477162
- [Derived] Kwon W, Hong D, Choi KH, Lee SH, Shin D, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Lee JM; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided Percutaneous Coronary Intervention Before and After Standardized Optimization Protocols. JACC Cardiovasc Interv. 2024 Jan 22;17(2):292-303. doi: 10.1016/j.jcin.2023.10.062. PMID 38267144
- [Derived] Kwon W, Choi KH, Song YB, Park YH, Lee JM, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Lee WS, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY; RENOVATE COMPLEX-PCI Investigators. Intravascular Imaging in Patients With Complex Coronary Lesions and Chronic Kidney Disease. JAMA Netw Open. 2023 Nov 1;6(11):e2345554. doi: 10.1001/jamanetworkopen.2023.45554. PMID 38019512
- [Derived] Kwon W, Lee JM, Yun KH, Choi KH, Lee SJ, Lee JY, Lee SY, Kim SM, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY, Song YB; RENOVATE COMPLEX-PCI Investigators. Clinical Benefit of Intravascular Imaging Compared With Conventional Angiography in Left Main Coronary Artery Intervention. Circ Cardiovasc Interv. 2023 Dec;16(12):e013359. doi: 10.1161/CIRCINTERVENTIONS.123.013359. Epub 2023 Nov 29. PMID 38018841
- [Derived] Lee JM, Choi KH, Song YB, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Jeong JO, Song PS, Doh JH, Jo SH, Yoon CH, Kang MG, Koh JS, Lee KY, Lim YH, Cho YH, Cho JM, Jang WJ, Chun KJ, Hong D, Park TK, Yang JH, Choi SH, Gwon HC, Hahn JY; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided or Angiography-Guided Complex PCI. N Engl J Med. 2023 May 4;388(18):1668-1679. doi: 10.1056/NEJMoa2216607. Epub 2023 Mar 5. PMID 36876735